CLINICAL TRIAL: NCT05660187
Title: Virtual Versus Usual In-office Care for Multiple Sclerosis: A Randomized Trial (VIRTUAL-MS)
Brief Title: VIRtual Versus UsuAL In-office Care for Multiple Sclerosis (VIRTUAL-MS)
Acronym: VIRTUAL-MS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: University of California, San Francisco (Other); University of Washington (Other)
Responsible Party: Principal Investigator, Marisa McGinley, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 23-045
Record Dates: First submitted 2022-12-13; First posted 2022-12-21 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-11

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; MS; telehealth; healthcare delivery
MeSH Terms: conditions — Multiple Sclerosis | interventions — Ambulatory Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telehealth care (Experimental): Telehealth visits will be performed using institutionally-approved, secure, web-based teleconferencing. The standard neurology visits will occur every 6 months with their established neurology clinician via telehealth. The comprehensive care will be offered via telehealth or within the patient's local community. The comprehensive care visits will be adapted for the individual participants' needs and symptoms, consistent with standard clinical care.
  Interventions: Other: Multiple Sclerosis Clinical Care Delivery via telehealth
- In-Clinic care (Active Comparator): Standard neurology visits will be conducted in-clinic visits every 6 months with their established neurology clinician. The comprehensive MS care visits will be conducted in-clinic. The comprehensive care visits will be adapted for the individual participants' needs and symptoms, consistent with standard clinical care.
  Interventions: Other: Multiple Sclerosis Clinical Care Delivery via standard in clinic visits

INTERVENTIONS:
Other: Multiple Sclerosis Clinical Care Delivery via telehealth — Intervention includes clinical care delivered via telehealth
  Arms: Telehealth care
Other: Multiple Sclerosis Clinical Care Delivery via standard in clinic visits — Intervention includes clinical care delivered via standard in clinic visits
  Arms: In-Clinic care

SUMMARY:
The current standard of outpatient MS care depends on in-clinic visits, but MS patients face many barriers to accessing this care. These barriers include those resulting from the disease itself, such as physical limitations, driving restrictions and financial limitations, and they are further compounded by an overall shortage of neurologists. Furthermore, MS care has a significant economic impact, with the estimated indirect and direct costs for treating MS in the US estimated to be > $85.4 billion. Therefore, there is a need to improve access to and reduce cost of MS care, and telehealth is a potential solution. The VIRTUAL-MS study has been designed to evaluate the impact of telehealth care on MS clinical outcomes, costs, and satisfaction compared to in-person care. Additionally, the study aims to evaluate facilitators and barriers to telehealth use to inform widespread implementation.

DETAILED DESCRIPTION:
The VIRTUAL-MS study aims to evaluate the impact of telehealth on MS care. The study will conduct a 24 month randomized controlled clinical trial at two Centers (Cleveland Clinic and University of California San Francisco) and will enroll 60 adult people with MS per Center with a recent diagnosis of MS. Participants will be randomized 1:1 to receive follow-up MS care via scheduled telehealth, or standard in-clinic, visits. All participants will have in-person visits at baseline and 24 months with in-person study visit including clinical assessments, patient reported outcomes, and medical history review. All participants will have clinical visits with their neurology clinician every 6 months (months 6, 12, and 18) via in-person or telehealth per randomized arm.

The primary objective of this study is to determine if MS care delivered via telehealth is non-inferior compared to in-clinic MS care as measured by worsening in one of the Multiple Sclerosis Functional Composite (MSFC) components at Month 24.

The secondary objectives of this study include the following:

* To determine if MS care delivered via telehealth has superior patient satisfaction compared to in-person MS care as measured by baseline to 24 month change in PSQ-18.
* To determine if MS care delivered via telehealth is more cost-effective than MS care delivered via in-person visits as measured by total non-medication costs over 24 months.

The researchers will also explore other clinical outcomes, treatment adherence, digital outcomes, patient experience, and clinician experience.

ELIGIBILITY:
Inclusion Criteria:

1. Ages ≥18
2. MS diagnosis within 24 months of randomization by 2017 McDonald Criteria.
3. Confirmatory MRI within 12 months prior to randomization.
4. Access to either mobile device, laptop or PC with internet connection to be able to conduct virtual visits
5. Participant's neurologist and/or advanced practice provider are participating in the study

Exclusion Criteria:

1. Clinically relevant condition that, in the opinion of the PI, could preclude participation in the study (e.g. neutropenia or wound care requiring frequent monitoring)
2. Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-03-31 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with disability progression | Baseline to 24 months
  The primary outcome will be disability worsening in one of the Multiple Sclerosis Functional Composite components at 24 months. Worsening is defined as 20% worsening in Timed 25 foot walking speed (T25FW), 20% worsening in the 9 hole peg test (9HPT), 20% worsening in Low Contrast Letter Acuity (LCLA) or a 4 point decrease in the Symbol Digit Modalities Test (SDMT).

SECONDARY OUTCOMES:
Change in Patient Satisfaction Questionnaire Short Form (PSQ-18) | Baseline to 24 months
  The secondary outcome will assess patient and clinical care team satisfaction via the Patient Satisfaction Questionnaire Short Form (PSQ-18) short form.
  Minimum value is 1 and maximum value is 5 for each question, where 5 means a better outcome.
Compare major healthcare costs | Baseline to 24 months
  The secondary outcome will compare major healthcare costs as measured by total non-medication costs.

CONTACTS AND LOCATIONS:
Overall Officials: Marisa McGinley, DO, Principal Investigator — The Cleveland Clinic; Riley Bove, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of California San Francisco, San Francisco, California
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McGinley M, Carlson JJ, Reihm J, Plow M, Roser M, Sisodia N, Cohen JA, Misra-Hebert AD, Lazar AA, Bove R. Virtual versus usual in-office care for multiple sclerosis: The VIRTUAL-MS multi-site randomized clinical trial study protocol. Contemp Clin Trials. 2024 Jul;142:107544. doi: 10.1016/j.cct.2024.107544. Epub 2024 Apr 23. PMID 38657731